CLINICAL TRIAL: NCT03365622
Title: Randomized, Double-Blind Clinical Study Evaluating Efficacy of Intravenous Versus Enteric Acetaminophen in Donor Nephrectomy and Robot-Assisted, Laparoscopic Nephrectomy.
Brief Title: Efficacy of IV Acetaminophen Versus Oral Acetaminophen
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Rochester (Other)
Responsible Party: Principal Investigator, Joseph W Dooley, MD, Associate Professor, University of Rochester
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 70162
Record Dates: First submitted 2017-11-30; First posted 2017-12-07 (Actual); Results first posted 2025-06-29 (Actual); Last update posted 2025-06-29 (Actual); Status verified 2025-06

CONDITIONS: Nephrectomy
MeSH Terms: interventions — Acetaminophen

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- IV acetaminophen and placebo pills (Active Comparator)
  Interventions: Drug: acetaminophen; Drug: Placebo Oral Tablet
- placebo IV (normal saline) + oral acetaminophen (Placebo Comparator)
  Interventions: Drug: Acetaminophen; Drug: Placebos

INTERVENTIONS:
Drug: acetaminophen — Active Intravenous doses will consist of a single 1,000mg/100 ml IV dose with contents of commercial vials transferred to an empty sterile IV bag.
  Arms: IV acetaminophen and placebo pills
Drug: Acetaminophen — 500mg acetaminophen tablet ,2 capsules oral every six hours for 24 hours
  Arms: placebo IV (normal saline) + oral acetaminophen
Drug: Placebos — Placebo Intravenous doses will consist of 100ml of normal saline transferred to an empty sterile IV bag.
  Arms: placebo IV (normal saline) + oral acetaminophen
Drug: Placebo Oral Tablet — Placebo, opaque capsules that have been filled with inert powder (lactose USP), 2 capsules oral every six hours for 24 hours
  Arms: IV acetaminophen and placebo pills

SUMMARY:
The aim of this study is to determine whether intravenous acetaminophen compared to enteric acetaminophen offers increased efficacy in patients who are scheduled for laparoscopic donor nephrectomy and for patients scheduled for robot-assisted, laparoscopic nephrectomy for cancer at the University of Rochester Medical Center. The standard surgical and post-operative care, including post-operative pain management will not be altered.

ELIGIBILITY:
Inclusion Criteria:

* Be at least 18 years old
* Be scheduled for donor nephrectomy or robot-assisted, laparoscopic nephrectomy for cancer at University of Rochester Medical Center
* Have cognitive ability to verbally rate their pain on the Numeric Rating Scale (NRS).

Exclusion Criteria:

* Age younger than 18 years old or older than 90 years old
* Pregnancy (Pre-operative pregnancy test is standard of care for all elective operating room cases)
* Weight less than 50 kg
* Epidural use
* History of known liver disease.
* Patient unable to take enteral medications.
* Be taking opioid medications chronically.

Ages: 18 Years to 89 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 214 (Actual)
Dates: Start 2018-08-08 (Actual); Primary Completion 2024-04-10 (Actual); Study Completion 2024-04-10 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- University of Rochester Medical Center, Rochester, New York, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Adult patients 18 years to 90 years old with the cognitive ability to rate their pain on the Numeric Rating Scale (NRS) and who were scheduled for laparoscopic donor nephrectomy, robot-assisted laparoscopic donor nephrectomy, or robot-assisted laparoscopic nephrectomy for renal cancer at the University of Rochester Medical Center (URMC) were eligible for enrollment.
Pre-assignment Details: There were 57 subjects who were withdrawn, however 6 of those subjects were included in the intent to treat analysis. as they did receive one dose of study medication.
Period: Overall Study
Arm/Group | IV Acetaminophen and Placebo Pills | Placebo IV (Normal Saline) + Oral Acetaminophen
Started | 108 | 106
Completed | 108 | 106
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | IV Acetaminophen and Placebo Pills | Placebo IV (Normal Saline) + Oral Acetaminophen | Total
Number analyzed (Participants) | 108 | 106 | 214
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 80 | 76 | 156
  >=65 years | 28 | 30 | 58
Age, Continuous [Mean (Standard Deviation); unit: Age in years] | 54.0 (14.6) | 54.4 (15.1) | 54.2 (14.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 51 | 58 | 109
  Male | 57 | 48 | 105
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 1
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 7 | 4 | 11
  White | 94 | 100 | 194
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 7 | 1 | 8
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 108 | 106 | 214
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 2 | 5
  Not Hispanic or Latino | 94 | 95 | 189
  Unknown or Not Reported | 11 | 9 | 20

OUTCOME MEASURES:

1. Primary Outcome: Total Opioid Dose (MME) Used in 24 Hours
Description: Total opiate dose used from the study start (when the first dose of acetaminophen is administered in the pre-anesthesia holding area) to 24 hours post-operatively (in morphine milligram equivalents (MME)).This will include opiates administered intra-operatively.
Time Frame: 20 to 24 hours post-operatively
Measure: Mean (Standard Deviation); unit: total morphine milligram equivalents
Arm/Group | IV Acetaminophen and Placebo Pills | Placebo IV (Normal Saline) + Oral Acetaminophen
Number analyzed (Participants) | 108 | 106
total morphine milligram equivalents | 103.61 (58.16) | 109.17 (57.59)
Statistical Analysis 1: Comparison: IV Acetaminophen and Placebo Pills vs Placebo IV (Normal Saline) + Oral Acetaminophen; A multiple linear regression model was used to examine the association between treatment assignment and the total opioid dose administered intraoperatively and postoperatively, adjusting for patient age, gender, body mass index (BMI), type of surgery (laparoscopic donor nephrectomy or laparoscopic nephrectomy for renal cancer), and whether the patient received a TAP block during surgery; Test type: Superiority; p = 0.3938, Regression, Linear; Adjusted for age, sex, BMI, type of surgery and TAP block; Mean Difference (Final Values) = 6.306, 95% CI 2-sided [-8.242 to 20.854], Standard Error of Mean 7.379 — The estimate reflects the adjusted difference in mean outcome between arms/groups, with the "placebo IV + oral acetaminophen" serving as the reference group

2. Secondary Outcome: Average Surgical Pain Intensity
Description: Average surgical pain intensity on a 0-10 numeric rating scale (NRS) administered between 20 and 24 hours post-operatively, with gatekeeping used to control for multiplicity. A larger NRS score means the patient is experiencing more pain, with 0 representing "no pain" and 10 representing "the worst possible pain".
Time Frame: 20-24 hours post-operatively
Population: A total of 6 participants were missing: 4 from the "IV acetaminophen" group and 2 from the "oral acetaminophen" group.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | IV Acetaminophen and Placebo Pills | Placebo IV (Normal Saline) + Oral Acetaminophen
Number analyzed (Participants) | 104 | 104
score on a scale | 4.87 (2.20) | 5.00 (1.96)
Statistical Analysis 1: Comparison: IV Acetaminophen and Placebo Pills vs Placebo IV (Normal Saline) + Oral Acetaminophen; A multiple linear regression model was used to examine the association between treatment assignment and the 20-24 hours post-op average surgical pain, adjusting for patient age, gender, body mass index (BMI), type of surgery (laparoscopic donor nephrectomy or laparoscopic nephrectomy for renal cancer), and whether the patient received a TAP block during surgery; Test type: Superiority; p = 0.7051, Regression, Linear; Adjusted for age, sex, BMI, type of surgery and TAP block; Mean Difference (Final Values) = 0.107, 95% CI 2-sided [-0.451 to 0.666], Standard Error of Mean 0.283 — [estimate comment as in outcome 1, analysis 1]

3. Secondary Outcome: Average Surgical Pain Intensity
Description: as for outcome 2
Time Frame: 1-2 hours post-operatively
Population: A total of 5 participants were missing: 3 from the "IV acetaminophen" group and 2 from the "oral acetaminophen" group.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | IV Acetaminophen and Placebo Pills | Placebo IV (Normal Saline) + Oral Acetaminophen
Number analyzed (Participants) | 105 | 104
score on a scale | 4.46 (2.34) | 4.77 (2.41)
Statistical Analysis 1: Comparison: IV Acetaminophen and Placebo Pills vs Placebo IV (Normal Saline) + Oral Acetaminophen; A multiple linear regression model was used to examine the association between treatment assignment and the 1-2 hours post-op average surgical pain, adjusting for patient age, gender, body mass index (BMI), type of surgery (laparoscopic donor nephrectomy or laparoscopic nephrectomy for renal cancer), and whether the patient received a TAP block during surgery; Test type: Superiority; p = 0.3852, Regression, Linear; Adjusted for age, sex, BMI, type of surgery and TAP block; Mean Difference (Final Values) = 0.276, 95% CI 2-sided [-0.349 to 0.901], Standard Error of Mean 0.317 — [estimate comment as in outcome 1, analysis 1]

4. Secondary Outcome: Mean Inspiratory Capacity
Description: The mean inspiratory capacity is presented as a percentage of the subject's baseline (pre-operative) inspiratory capacity, recorded at the time of pain intensity assessments between 1-2 hours postoperatively. Inspiratory capacity is measured using a Voldyne 5000 incentive spirometer (Hudson RCI, Teleflex Medical) and recorded in milliliters to the nearest 250 cc mark on the incentive spirometer. Higher percentages reflect better recovery of inspiratory function.
Time Frame: 1-2 hours post-operatively
Population: A total of 6 participants were missing: 3 from the "IV acetaminophen" group and 3 from the "oral acetaminophen" group.
Measure: Mean (Standard Deviation); unit: percent of baseline inspiratory capacity
Arm/Group | IV Acetaminophen and Placebo Pills | Placebo IV (Normal Saline) + Oral Acetaminophen
Number analyzed (Participants) | 105 | 103
percent of baseline inspiratory capacity | 66.60 (20.26) | 67.07 (20.74)
Statistical Analysis 1: Comparison: IV Acetaminophen and Placebo Pills vs Placebo IV (Normal Saline) + Oral Acetaminophen; A multiple linear regression model was used to examine the association between treatment assignment and the 1-2 hours post-op inspiratory capacity percentage, adjusting for patient age, gender, body mass index (BMI), type of surgery (laparoscopic donor nephrectomy or laparoscopic nephrectomy for renal cancer), and whether the patient received a TAP block during surgery; Test type: Superiority; p = 0.8498, Regression, Linear; Adjusted for age, sex, BMI, type of surgery and TAP block; Mean Difference (Final Values) = 0.534, 95% CI 2-sided [-5.02 to 6.088], Standard Error of Mean 2.816 — [estimate comment as in outcome 1, analysis 1]

5. Secondary Outcome: Mean Inspiratory Capacity
Description: The mean inspiratory capacity is presented as a percentage of the subject's baseline (pre-operative) inspiratory capacity, recorded at the time of pain intensity assessments between 20-24 hours postoperatively. Inspiratory capacity is measured using a Voldyne 5000 incentive spirometer (Hudson RCI, Teleflex Medical) and recorded in milliliters to the nearest 250 cc mark on the incentive spirometer. Higher percentages reflect better recovery of inspiratory function.
Time Frame: 20-24 hours post-operatively
Population: A total of 7 participants were missing: 4 from the "IV acetaminophen" group and 3 from the "oral acetaminophen" group.
Measure: Mean (Standard Deviation); unit: percent of baseline inspiratory capacity
Arm/Group | IV Acetaminophen and Placebo Pills | Placebo IV (Normal Saline) + Oral Acetaminophen
Number analyzed (Participants) | 104 | 103
percent of baseline inspiratory capacity | 64.41 (21.82) | 63.35 (22.57)
Statistical Analysis 1: Comparison: IV Acetaminophen and Placebo Pills vs Placebo IV (Normal Saline) + Oral Acetaminophen; A multiple linear regression model was used to examine the association between treatment assignment and the 20-24 hours post-op inspiratory capacity percentage, adjusting for patient age, gender, body mass index (BMI), type of surgery (laparoscopic donor nephrectomy or laparoscopic nephrectomy for renal cancer), and whether the patient received a TAP block during surgery; Test type: Superiority; p = 0.5839, Regression, Linear; Adjusted for age, sex, BMI, type of surgery and TAP block; Mean Difference (Final Values) = -1.650, 95% CI 2-sided [-7.579 to 4.28], Standard Error of Mean 3.007 — [estimate comment as in outcome 1, analysis 1]

6. Secondary Outcome: Dynamic Pain Score During Incentive Spirometer Use
Description: Dynamic pain score on a 0-10 numeric rating scale (NRS) with incentive spirometer use taken during pain intensity assessments at 1-2 hours post-operatively. A larger NRS score means the patient is experiencing more pain, with 0 representing "no pain" and 10 representing "the worst possible pain".
Time Frame: 1-2 hours post-operatively
Population: A total of 6 participants were missing: 3 from the "IV acetaminophen" group and 3 from the "oral acetaminophen" group.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | IV Acetaminophen and Placebo Pills | Placebo IV (Normal Saline) + Oral Acetaminophen
Number analyzed (Participants) | 105 | 103
score on a scale | 4.73 (2.71) | 5.15 (2.51)
Statistical Analysis 1: Comparison: IV Acetaminophen and Placebo Pills vs Placebo IV (Normal Saline) + Oral Acetaminophen; A multiple linear regression model was used to examine the association between treatment assignment and the 1-2 hours post-op dynamic pain score, adjusting for patient age, gender, body mass index (BMI), type of surgery (laparoscopic donor nephrectomy or laparoscopic nephrectomy for renal cancer), and whether the patient received a TAP block during surgery; Test type: Superiority; p = 0.2479, Regression, Linear; Adjusted for age, sex, BMI, type of surgery and TAP block; Mean Difference (Final Values) = 0.399, 95% CI 2-sided [-0.280 to 1.078], Standard Error of Mean 0.344 — [estimate comment as in outcome 1, analysis 1]

7. Secondary Outcome: Dynamic Pain Score During Incentive Spirometer Use
Description: Dynamic pain score on a 0-10 numeric rating scale (NRS) with incentive spirometer use taken during pain intensity assessments at 20-24 hours post-operatively. A larger NRS score means the patient is experiencing more pain, with 0 representing "no pain" and 10 representing "the worst possible pain".
Time Frame: 20-24 hours post-operatively
Population: A total of 9 participants were missing: 5 from the "IV acetaminophen" group and 4 from the "oral acetaminophen" group.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | IV Acetaminophen and Placebo Pills | Placebo IV (Normal Saline) + Oral Acetaminophen
Number analyzed (Participants) | 103 | 102
score on a scale | 4.62 (2.56) | 5.12 (2.25)
Statistical Analysis 1: Comparison: IV Acetaminophen and Placebo Pills vs Placebo IV (Normal Saline) + Oral Acetaminophen; A multiple linear regression model was used to examine the association between treatment assignment and the 20-24 hours post-op dynamic pain score, adjusting for patient age, gender, body mass index (BMI), type of surgery (laparoscopic donor nephrectomy or laparoscopic nephrectomy for renal cancer), and whether the patient received a TAP block during surgery; Test type: Superiority; p = 0.1502, Regression, Linear; Adjusted for age, sex, BMI, type of surgery and TAP block; Mean Difference (Final Values) = 0.484, 95% CI 2-sided [-0.177 to 1.145], Standard Error of Mean 0.335 — [estimate comment as in outcome 1, analysis 1]

8. Secondary Outcome: Surgical Pain Score During the 20-24 Hour Assessment
Description: Pain intensity on a 0-10 numeric rating scale (NRS) prior to incentive spirometry use was taken during pain intensity assessments at 20-24 hours post-operatively. A larger NRS score means the patient is experiencing more pain, with 0 representing "no pain" and 10 representing "the worst possible pain".
Time Frame: 20-24 hours post-operatively
Population: A total of 16 participants were missing: 10 from the "IV acetaminophen" group and 6 from the "oral acetaminophen" group.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | IV Acetaminophen and Placebo Pills | Placebo IV (Normal Saline) + Oral Acetaminophen
Number analyzed (Participants) | 98 | 100
score on a scale | 3.52 (2.25) | 3.89 (2.14)
Statistical Analysis 1: Comparison: IV Acetaminophen and Placebo Pills vs Placebo IV (Normal Saline) + Oral Acetaminophen; A multiple linear regression model was used to examine the association between treatment assignment and the 20-24 hours post-op surgical pain score, adjusting for patient age, gender, body mass index (BMI), type of surgery (laparoscopic donor nephrectomy or laparoscopic nephrectomy for renal cancer), and whether the patient received a TAP block during surgery; Test type: Superiority; p = 0.2797, Regression, Linear; Adjusted for age, sex, BMI, type of surgery and TAP block; Mean Difference (Final Values) = 0.339, 95% CI 2-sided [-0.278 to 0.955], Standard Error of Mean 0.313 — [estimate comment as in outcome 1, analysis 1]

9. Secondary Outcome: Time to First Narcotic Use
Description: Time to first postoperative narcotic use, measured in hours (range: 1 to 24).
Time Frame: 24 hours post-operatively
Population: A total of 24 participants were missing: 14 from the "IV acetaminophen" group and 10 from the "oral acetaminophen" group.
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | IV Acetaminophen and Placebo Pills | Placebo IV (Normal Saline) + Oral Acetaminophen
Number analyzed (Participants) | 94 | 96
hours | 3.31 (5.34) | 2.85 (4.91)
Statistical Analysis 1: Comparison: IV Acetaminophen and Placebo Pills vs Placebo IV (Normal Saline) + Oral Acetaminophen; A multiple linear regression model was used to examine the association between treatment assignment and time to first narcotic use, adjusting for patient age, gender, body mass index (BMI), type of surgery (laparoscopic donor nephrectomy or laparoscopic nephrectomy for renal cancer), and whether the patient received a TAP block during surgery; Test type: Superiority; p = 0.6527, Regression, Linear; Adjusted for age, sex, BMI, type of surgery and TAP block; Mean Difference (Final Values) = -0.333, 95% CI 2-sided [-1.792 to 1.125], Standard Error of Mean 0.739 — [estimate comment as in outcome 1, analysis 1]

10. Secondary Outcome: Number of Participants With Nausea
Description: Number of participants with nausea was assessed based on the administration of anti-emetic medications, with a value of 0 indicating no nausea and 1 indicating the presence of nausea.
Time Frame: 24 hours post-operatively
Measure: Count of Participants; unit: Participants
Arm/Group | IV Acetaminophen and Placebo Pills | Placebo IV (Normal Saline) + Oral Acetaminophen
Number analyzed (Participants) | 108 | 106
Participants | 58 | 40
Statistical Analysis 1: Comparison: IV Acetaminophen and Placebo Pills vs Placebo IV (Normal Saline) + Oral Acetaminophen; A logistic regression model was used to examine the association between treatment assignment and incidence of nausea, adjusting for patient age, gender, body mass index (BMI), type of surgery (laparoscopic donor nephrectomy or laparoscopic nephrectomy for renal cancer), and whether the patient received a TAP block during surgery; Test type: Superiority; p = 0.0499, Regression, Logistic; Adjusted for age, sex, BMI, type of surgery and TAP block; Odds Ratio (OR) = 0.465, 95% CI 2-sided [0.217 to 1.000]

11. Secondary Outcome: Time to Discharge From Post-anesthesia Care Unit
Description: Length of time in minutes from PACU(post-anesthesia care unit) arrival to discharge.
Time Frame: 24 hours
Measure: Mean (Standard Deviation); unit: Minutes
Arm/Group | IV Acetaminophen and Placebo Pills | Placebo IV (Normal Saline) + Oral Acetaminophen
Number analyzed (Participants) | 108 | 106
Minutes | 174.17 (82.99) | 195.48 (170.41)
Statistical Analysis 1: Comparison: IV Acetaminophen and Placebo Pills vs Placebo IV (Normal Saline) + Oral Acetaminophen; A multiple linear regression model was used to examine the association between treatment assignment and time to discharge from PACU, adjusting for patient age, gender, body mass index (BMI), type of surgery (laparoscopic donor nephrectomy or laparoscopic nephrectomy for renal cancer), and whether the patient received a TAP block during surgery; Test type: Superiority; p = 0.179, Regression, Linear; Adjusted for age, sex, BMI, type of surgery and TAP block; Mean Difference (Final Values) = 24.492, 95% CI 2-sided [-11.321 to 60.304], Standard Error of Mean 18.165 — [estimate comment as in outcome 1, analysis 1]

12. Secondary Outcome: Time to Hospital Discharge
Description: Number of days to discharge from hospital
Time Frame: 30 days
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | IV Acetaminophen and Placebo Pills | Placebo IV (Normal Saline) + Oral Acetaminophen
Number analyzed (Participants) | 108 | 106
Days | 2.33 (1.30) | 2.60 (2.27)
Statistical Analysis 1: Comparison: IV Acetaminophen and Placebo Pills vs Placebo IV (Normal Saline) + Oral Acetaminophen; A multiple linear regression model was used to examine the association between treatment assignment and time to hospital discharge, adjusting for patient age, gender, body mass index (BMI), type of surgery (laparoscopic donor nephrectomy or laparoscopic nephrectomy for renal cancer), and whether the patient received a TAP block during surgery; Test type: Superiority; p = 0.2811, Regression, Linear; Adjusted for age, sex, BMI, type of surgery and TAP block; Mean Difference (Final Values) = 0.274, 95% CI 2-sided [-0.226 to 0.773], Standard Error of Mean 0.253 — [estimate comment as in outcome 1, analysis 1]

ADVERSE EVENTS:
Time Frame: Up to 24 hours post-operatively or until hospital discharge
Arm/Group | IV Acetaminophen and Placebo Pills | Placebo IV (Normal Saline) + Oral Acetaminophen
All-Cause Mortality (participants affected / at risk) | 0/108 | 0/106
Serious Adverse Events (participants affected / at risk) | 1/108 | 1/106
Other Adverse Events (participants affected / at risk) | 14/108 | 16/106
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | IV Acetaminophen and Placebo Pills (N=108) | Placebo IV (Normal Saline) + Oral Acetaminophen (N=106)
Anemias non-hemolytic and marrow depression (Blood and lymphatic system disorders) | 1 | 0
Cognitive and attention disorders (Nervous system disorders) | 0 | 1
Urinary tract infections and Epididymal and testicular infections (Infections and infestations) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | IV Acetaminophen and Placebo Pills (N=108) | Placebo IV (Normal Saline) + Oral Acetaminophen (N=106)
Gastrointestinal symptoms (Gastrointestinal disorders) | 2 | 2
Anemias non-hemolytic and marrow depression (Blood and lymphatic system disorders) | 1 | 1
Corneal disorders (Eye disorders) | 2 | 0
Respiratory failures and dysfunctions (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Muscle disorders (Musculoskeletal and connective tissue disorders) | 0 | 2
Joint disorders (Musculoskeletal and connective tissue disorders) | 2 | 2
Intraoperative and post-op hemorrhages (Vascular disorders) | 2 | 0
Cardiac arrhythmias (Cardiac disorders) | 0 | 1
Liver function analyses (Hepatobiliary disorders) | 1 | 0
Air leak syndromes (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Body temperature conditions (General disorders) | 0 | 1
Renal function analyses (Renal and urinary disorders) | 0 | 1
Infusion site reactions (General disorders) | 0 | 1
Vascular hypotensive disorders (Vascular disorders) | 1 | 0
Hypotension post-op (Vascular disorders) | 0 | 1
Systemic and deep-seated mycoses (Infections and infestations) | 0 | 1
Post-op disorder of lymphatic vessels (Blood and lymphatic system disorders) | 1 | 0
Renal function analyses & White blook cell abnormal (Renal and urinary disorders) | 0 | 1
Skin ulcerations and conditions necrotic (Skin and subcutaneous tissue disorders) | 0 | 1
Peripheral neuropathies (Nervous system disorders) | 0 | 1
Respiratory failure post-op (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Postoperative ileus (Gastrointestinal disorders) | 0 | 1
Acute and chronic renal failures (Renal and urinary disorders) | 0 | 1
Abnormal kidney function analyses (Renal and urinary disorders) | 1 | 0
Electrolyte and fluid balance conditions (Metabolism and nutrition disorders) | 1 | 0

LIMITATIONS AND CAVEATS:
The main limitation was the addition of TAP blocks mid-study for laparoscopic nephrectomy patients. This change likely didn't affect results, as both groups had similar exposure. Variability in gastric drainage, delayed PACU dosing due to lethargy, and prolonged procedures may have influenced outcomes. Lastly, no control group without acetaminophen was included due to ethical concerns over withholding standard pain management.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2023-01-13): https://cdn.clinicaltrials.gov/large-docs/22/NCT03365622/Prot_SAP_000.pdf
  • Informed Consent Form (2023-01-13): https://cdn.clinicaltrials.gov/large-docs/22/NCT03365622/ICF_001.pdf